CLINICAL TRIAL: NCT05514652
Title: Development of Anesthesia Standard Operating Procedure During On-pump Coronary Artery Bypass Grafting Due to Coronary Heart Disease
Brief Title: Anesthesia Standard Operating Procedure During On-pump Coronary Artery Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heart Institute, Ministry of Health of Ukraine (Other)
Responsible Party: Principal Investigator, Maruniak Stepan, Senior Researcher, Heart Institute, Ministry of Health of Ukraine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180001
Record Dates: First submitted 2022-08-19; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease; Low Cardiac Output Syndrome; Atrial Fibrillation; Postoperative Complications
Keywords: coronary artery bypass grafting; cardiopulmonary bypass; coronary artery disease; low cardiac output syndrome; low-dose opioid anesthesia; postoperarive atrial fibrillation; IL-6
MeSH Terms: conditions — Coronary Artery Disease; Cardiac Output, Low; Atrial Fibrillation; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Experimental): Multimodal low-opioid protocol provided for induction of anesthesia with intravenous (iv) propofol administration using the dosage of 1.5-2 mg/kg at 40 mg in interval of 10-15 seconds, iv fentanyl dosage 1-1.5 μg/kg and iv pipecuronium bromide dosage of 0.1 mg/kg. Before intubation of the trachea, a lidocaine 1 mg / kg bolus was added intravenously, with the simultaneous establishment of a continuous infusion at a dose of 1.5-2 mg/kg/h. All patients were administered a bolus of ketamine (0.5 mg/kg) and were started continuous infusion dexmedetomidine at a dose 0.7 μg/kg/h. If indicated fentanyl was used as additional analgesic during surgery by bolus injection. Depth of anesthesia was monitored with bispectral index; the dosage of sevoflurane from 1,5vol% to 2,5vol% was titrated to maintain BIS values from 40 to 60.
  Interventions: Drug: Low opioid anesthesia
- Second group (Active Comparator): Routine opioid protocol of anesthesia provided for induction of anesthesia with the iv administration of propofol dosage of 1.5-2 mg/kg at 40 mg in interval of 15-20 seconds, iv fentanyl at a dose of 1-1.5 μg/kg and iv pipecuronium bromide dosage of 0.1 mg/kg. For analgesia, bolus injections of fentanyl were used at a dose of 8-10 μg/kg for the entire duration of the operation, muscle relaxation - pipecuronium bromide at a dose of 0.1 mg/kg. Depth of anesthesia was monitored with bispectral index; the dosage of sevoflurane from 1,5vol% to 2,5vol% was titrated to maintain BIS values from 40 to 60.
  Interventions: Drug: Low opioid anesthesia

INTERVENTIONS:
Drug: Low opioid anesthesia — Multimodal low-dose opioid protocol for anesthesia based on ketamine, lidocaine and dexmedetomidine

SUMMARY:
Background: Despite improvements in surgical and anesthesia procedures over the past 15 years complications during cardiac surgery still remain high. Bridgewater B et al. describes mortality during on-pump coronary artery bypass grafting (CABG) at 2%-3%, and the rate postoperative complications about 20%-30%. At the same time, the standard of care in patients undergoingon-pump CABG is not fully established.

Hypothesis, Research Need: Use of multimodal low-dose opioid anesthesia during CABG decreases inflammatory response and the incidence of early postoperative cardiac complications due to a reduction in interleukin-6.

Methodology: According to anesthesia standard protocol, all patients were divided into two groups - study group with multimodal low-dose opioid anesthesia (60 patients) and control group with a high-dose opioid anesthesia (60 patients). Primary (IL-6 at the end of the operation) and secondary clinical outcomes (postoperative atrial fibrillation (POAF), low cardiac output syndrome (LCOS), duration of mechanical ventilation (MV), length of intensive care unit (ICU) stay, length of hospital stay) were compared between the groups.

Analysis Tools: Clinical observations; instrumental research methods (electrocapdiography, echocardiography); labs (blood gases, hemoglobin, electrolytes); enzyme-linked immunosorbent assay (IL-6); statistical (Student's t-test, Mann-Whitney U test, χ2-test, correlation analysis).

Expected Outcomes: Use of multimodal low-dose opioid anesthesia during CABG will decrease inflammatory response (lower levels of IL-6 at the end of the surgery) and the incidence of early postoperative cardiac complications, expressed as lower incidence of LCOS and POAF, lower duration of MV and lower length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* age from 44 to 65 years,
* nn ejection fraction > 30%,
* operational risk assessment for EuroSCORE II <5%,
* on-pump coronary artery bypass grafting

Exclusion Criteria:

* patient's refusal
* off-pump coronary artery bypass grafting
* the need for additional intervention on the heart

Ages: 44 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of concentration of IL-6 in venous blood plasma immediately after the surgery | immediately after surgery
Number of people with low cardiac output syndrome | immediately after the surgery
  Postoperative low cardiac output syndrome (LCOS) was defined as hemodynamic instability requiring continued pharmacologic support with 2 inotropic medications (epinephrine, milrinone, dobutamine) on postoperative day 1
Number of people with postoperative atrial fibrillation | immediately after the surgery
  Postoperative atrial fibrillation was defined as first appeared in the period immediately after surgery
Duration of mechanical ventilation | immediately after the surgery
  The decision about the extubation was made on the basis of following clinical criteria: recovering from muscle relaxation and anesthesia; patients is easy to rouse, neurologically intact, lift head and sticks out tongue; stable hemodynamics (heart rate and blood pressure are within ordered parameters, bleeding is controlled); spontaneous muscle movement with stable respiratory rate and adequate oxygenation, which was confirmed by arterial blood gases (SaO2 >92 %, on FiO2 <50%).
The length of ICU stay | immediately after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute Ministry of Health of Ukraine, Kyiv, Kyiv Regio, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stepan M, Oleh L, Oleksandr D, Justyna S. Effects of multimodal low-opioid anesthesia protocol during on-pump coronary artery bypass grafting: a prospective cohort study. J Cardiothorac Surg. 2023 Oct 6;18(1):272. doi: 10.1186/s13019-023-02395-y. PMID 37803334